CLINICAL TRIAL: NCT05980338
Title: Comparative Study Between Knee Genicular Nerve Ablation by Thermal Radiofrequency vs Thermal Radiofrequency Plus Alcohol Neurolysis for Treatment of Symptomatic Knee Osteoarthritis
Brief Title: Knee Genicular Nerve Ablation by Thermal Radiofrequency vs Thermal Radiofrequency Plus Alcohol Neurolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Lydia edward aziz zakhary, Principal Investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: knee genicular nerve ablation
Record Dates: First submitted 2023-07-08; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): The patients are placed in supine position with knee preparation using an iodine-based product and drape in a sterile manner Then the ground pad of the radio frequency machine will be placed in the other leg (we used the Neurotherm NT1100 re generator) All the patients will be monitored by ECG, noninvasive blood pressure and pulse oximetry The 3 entry sites will be detected under fluoroscopy then local anesthesia will be performed using lidocaine 2% followed by the insertion of the 3 radiofrequency cannulas (STRYKER 20 G, 9 cm with 1 cm active tip) targeting the 3 main nerves ( superior medial genicular, superior lateral genicular and the inferior medial genicular nerves ). this group will receive radio frequency alone .
  Interventions: Procedure: genicular nerve ablation by thermal radiofrequency
- study group (Experimental): this group will pass through the all steps but after the radiofrequency is done at each level a 1 ml of 70% alcohol will be injected making a total of 3 ml injection to each nerve.
  Interventions: Procedure: genicular nerve ablation by thermal radiofrequency; Procedure: genicular nerve ablation by thermal radiofrequency plus alcohol neurolysis

INTERVENTIONS:
Procedure: genicular nerve ablation by thermal radiofrequency — radio-frequency will be done using the Neurotherm NT1100 re-generator. The 3 entry sites will be detected under fluoroscopy then local anesthesia will be performed using lidocaine 2% followed by the insertion of the 3 radiofrequency cannulas (STRYKER 20 G, 9 cm with 1 cm active tip) targeting the 3 main nerves ( superior medial genicular, superior lateral genicular and the inferior medial genicular nerves ) .
  A confirmation of the targeted sites is done under fluoroscopy in both A-P and lateral views then a motor stimulation will be done to ensure no undesirable motor response followed by lidocaine 1 % injection and placing of the radiofrequency cables and ablation was done at 80 degrees for 90 seconds . The procedure will be repeated 3 times at different levels in the lateral view separated by 0,5 cm to ensure successful targeting. Then remove the needles.
Procedure: genicular nerve ablation by thermal radiofrequency plus alcohol neurolysis — radio-frequency will be done using the Neurotherm NT1100 re-generator. The 3 entry sites will be detected under fluoroscopy then local anesthesia will be performed using lidocaine 2% followed by the insertion of the 3 radiofrequency cannulas (STRYKER 20 G, 9 cm with 1 cm active tip) targeting the 3 main nerves of the knee.
  A confirmation of the targeted sites is done under fluoroscopy in both A-P and lateral views then a motor stimulation will be done to ensure no undesirable motor response followed by lidocaine 1 % injection and placing of the radio-frequency cables and ablation was done at 80 degrees for 90 seconds . The procedure will be repeated 3 times at different levels in the lateral view. After the radiofrequency is done at each level a 1 ml of 70% alcohol will be injected making a total of 3 ml injection to each nerve Then remove the needles.
  Arms: study group

SUMMARY:
the aim of our study is to compare effectiveness (satisfaction) and duration of pain relief between patients receiving the conventional thermal radiofrequency on the genicular nerves alone vs patients who will receive the conventional method plus alcohol neurolysis of the targeted nerves.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders.
2. Age between 60-70 years.
3. ASA 1,2 & 3 physical status.
4. x ray imaging confirming the osteoarthritis and unwell or not candidate for knee replacement surgery

Exclusion Criteria:

1. Neurological disorders.(previous cerebrovascular stroke , neuropathy , or weakness )
2. coagulopathy ( plt < 50000, INR > 1.7 )
3. Infection at or near the injection site.
4. presence of pacemaker or defibrillator 5 - Acute knee injury.

6- age < 60 or >70 years

Ages: 60 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2023-06-17 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
pain relief after 1 month | 1 month
  evaluating degree of pain relief after knee genicular nerve ablation by thermal radiofrequency plus alcohol neurolysis using numeric pain rating scale ( 11 number score scale where 0 indicates no pain and 10 indicates worst pain imaginable )after 1 month.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Kidd VD, Strum SR, Strum DS, Shah J. Genicular Nerve Radiofrequency Ablation for Painful Knee Arthritis: The Why and the How. JBJS Essent Surg Tech. 2019 Mar 13;9(1):e10. doi: 10.2106/JBJS.ST.18.00016. eCollection 2019 Mar 26. PMID 31333900
- [Background] Liu J, Wang T, Zhu ZH. Efficacy and safety of radiofrequency treatment for improving knee pain and function in knee osteoarthritis: a meta-analysis of randomized controlled trials. J Orthop Surg Res. 2022 Jan 15;17(1):21. doi: 10.1186/s13018-021-02906-4. PMID 35033150
- [Background] Dass RM, Kim E, Kim HK, Lee JY, Lee HJ, Rhee SJ. Alcohol neurolysis of genicular nerve for chronic knee pain. Korean J Pain. 2019 Jul 1;32(3):223-227. doi: 10.3344/kjp.2019.32.3.223. PMID 31257831